CLINICAL TRIAL: NCT01421771
Title: Blood Pressure in Dialysis Patients (BID Study)
Brief Title: Blood Pressure in Dialysis Patients
Acronym: BID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Tufts Medical Center (Other); Medical University of South Carolina (Other); University of Pittsburgh Medical Center (Other); The Cleveland Clinic (Other); Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DK083424-01A1 (NIH)
Record Dates: First submitted 2011-08-16; First posted 2011-08-23 (Estimated); Results first posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Hypertension; Renal Failure Chronic Requiring Hemodialysis; Blood Pressure; Dialysis
MeSH Terms: conditions — Hypertension | interventions — Antihypertensive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment to an intensive BP goal (Active Comparator): Treatment to a pre-dialysis standardized dialysis unit systolic blood pressure of 110-140 mm Hg
  Interventions: Drug: Antihypertensive Agents; Other: Dry weight Challenge; Dietary Supplement: Extend dialysis treatment time and re-challenge estimated dry weight
- Treatment to standard BP goal (Placebo Comparator): Treatment to a pre-dialysis Standardized dialysis unit systolic BP of 155-165 mm Hg
  Interventions: Drug: Antihypertensive Agents; Other: Dry weight Challenge; Dietary Supplement: Extend dialysis treatment time and re-challenge estimated dry weight

INTERVENTIONS:
Drug: Antihypertensive Agents — Study formulary consists of ACE/ARB, Beta Adrenergic Blocker, Calcium Channel Blocker, vasodilators, peripheral alpha antagonist and central alpha agonist.
  ACE I or ARB is first line, the order of addition of subsequent medications is per the discretion of the investigator
Other: Dry weight Challenge — Reduce the estimated dry weight of the patient's progressively over 2 -week intervals until the dry weight challenge is no longer tolerated or the patient is at BP goal
Dietary Supplement: Extend dialysis treatment time and re-challenge estimated dry weight — Extend dialysis treatment time and re-challenge estimated dry weight

SUMMARY:
Hypertension is a major cause of cardiovascular (CV) morbidity and mortality. Although studies in the general population have demonstrated a continuous reduction in CV risk with each mmHg drop in systolic blood pressure (SBP), multiple observational studies conducted in hemodialysis (HD) patients have demonstrated that patients with mild to moderate hypertension may have decreased mortality compared to those with normal blood pressure (BP). The investigators recently reported that among HD patients, those with routine pre-dialysis BP values that met the Kidney Disease Outcomes Quality Initiative (KDOQI) guidelines (<140/90 mm Hg) had increased mortality compared to patients with mild to moderate hypertension. However, these observational studies included untreated patients in whom low or normal BP may reflect significant cardiac disease or other comorbid conditions. In the setting of reduced vascular compliance and impaired autoregulation, aggressive BP lowering may decrease coronary or cerebral perfusion. Thus, it is unclear if aggressive BP lowering will be harmful or beneficial. A well-designed randomized control trial (RCT) is needed to answer this important question. Prior to conducting a full-scale RCT it is prudent to conduct a pilot study to assess feasibility and inform the design of the former. The investigators propose to conduct a pilot RCT in a prevalent cohort of HD patients to assess the safety and feasibility of treating patients to a low (110-140 mmHg)and standard (155-165) mm Hg pre-dialysis BP target.

DETAILED DESCRIPTION:
Mortality and morbidity among hemodialysis (HD) patients remain unacceptably high, thus there is a compelling need to improve clinical outcomes. Accordingly, the National Kidney Foundation's Kidney Disease Outcome Quality Improvement program (KDOQI) has published a guideline calling for a pre-dialysis systolic blood pressure (SBP) <140 mmHg in HD patients. However, the evidence supporting this guideline was graded as weak since it was largely extrapolated from the general population. Studies in the general population have demonstrated a continuous reduction in cardiovascular risk with each mmHg drop in systolic blood pressure (SBP), extending below levels that were in past considered "normal". The Systolic Blood Pressure Intervention Trial (SPRINT) study has showed a decrease in the composite outcome of CV events and CV mortality among non-diabetic patients at high risk for cardiovascular events by targeting a SBP of <120 mmHg. It is reasonable to postulate that intensive control of BP may be beneficial in HD patients, who in many ways resemble patients in SPRINT except that they have progressed to end stage renal disease. Thus, it is timely to propose conducting a RCT of intensive versus standard control of blood pressure in HD patients.

The investigators recognize that from observational studies suggest that mortality among HD patients may be increased among patients who meet the current KDOQI guideline. Unidentified confounders may have contributed to these surprising findings. The conclusions reached by observational studies in HD patients have often been refuted by randomized controlled trials (RCTs). Therefore, a RCT is needed to determine if a pre-dialysis SBP <140 mmHg specified by KDOQI is an appropriate target. Prior to beginning a full-scale-RCT, it is imperative to conduct a pilot study to demonstrate safety and efficacy and to inform the design of the full-scale study. The pilot study is designed to answer the following questions:

1. What are the estimated recruitment, accrual and retention rates?
2. What proportions of patients in each arm will achieve and maintain SBP within the assigned target and will the investigators achieve equal or greater than 10mmHg separation in the average SBP between the two arms?
3. What are the anticipated adverse and serious adverse events rates within the intensive and standard arms?
4. What end points should be used in the full-scale trial?
5. What blood pressure (BP) measurements e.g., routine dialysis unit BP (RDUBPM), standardized dialysis unit BP (SDUBPM), standardized home BP (HBPM) or ambulatory BP monitoring (ABPM) to guide therapy? Although SDUBPM, HBPM and ABPM may be more powerful than RDUBP in predicting clinical outcomes,long term adherence with these techniques has not been demonstrated.

Specific Aims

1. Establish procedures for SDUBPM, HBPM and ABPM and web-based data entry.
2. Recruit and randomize patients into two treatment arms with target pre-dialysis SDUSBPM values <140 and < 160 mmHg and measure recruitment, accrual, and dropout rates in each arm.
3. Assess the feasibility of attaining and maintaining these targets and the degree of SBP separation achieved during a one year intervention.
4. Measure adherence rates for obtaining protocol SDUBPM, HBPM and ABPM over the one-year intervention.
5. Assess the safety of treating participants to the study's SBP targets by measuring occurrence rates of CVD and non-CVD morbidity and mortality and other adverse and serious adverse events in each arm.
6. Compare the differences in changes in left ventricular mass index (LVMI), aortic pulse wave velocity(APWV), and aortic distensibility, respectively, between the two study arms.
7. Conduct statistical analyses to inform the design of the full-scale study.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years
2. On thrice weekly maintenance hemodialysis for greater than 90 days
3. For entry into baseline period: 2-week average RDUSBPM > 155 mm Hg on AHT medications or < 155 mm Hg on ≥ 1 AHT medications For randomization: 2-week average SDUSBPM ≥ 155 mm Hg

Exclusion Criteria:

1. Two- week average, pre-dialysis mid-week SDUSBPM ≥180 mmHg on maximal doses of ≥ 4 antihypertensive agents;
2. Inability to measure blood pressures in an upper arm;
3. History of inter or post-dialytic hypotension (defined as systolic blood pressure <90 mmHg) within the past 2 weeks or inter- or post- dialytic hypotension requiring hospitalization (including emergency room visit) and/or the use of midodrine in the past 6 months;
4. Required one or more urgent, unscheduled dialysis treatment for congestive heart failure in the past 3 months (other than in an incident patient at the time of starting dialysis);
5. Acute myocardial infarction, unstable angina or stroke/ TIA in past three the 3 months;
6. Severe aortic valve stenosis (valve area <1cm 2) carotid artery stenosis (>70% stenosis);
7. Known abdominal aortic aneurysm >5 cm in diameter or thoracic aortic aneurysm of any diameter;
8. Body mass index >40 kg/m2 or arm circumference > 52 cm, which precludes measuring blood pressure with the "thigh" blood pressure cuff;
9. Life expectancy <1 year;
10. A living donor, kidney transplant, or switch to peritoneal dialysis scheduled within the next year;
11. Significant cognitive impairment;
12. spKt/V ≤1.2 in the past 2 months;
13. Active liver disease;
14. Active alcohol or substance abuse including narcotics within the past year;
15. Contraindication to cardiac MRI;
16. Current or planned pregnancy within the next year;
17. Unwillingness to consent to pregnancy test and/or use of birth control if of childbearing potential;
18. Suspicion that the participant will not be willing or able to adhere to prescribed medications and study protocol;
19. Incarcerated;
20. Significant concern about the study expressed by spouse, significant other, family member primary nephrologist or primary care physician;
21. Participation in another intervention study;
22. Unable to speak or understand English or Spanish;
23. Plan to relocate within one year;
24. participation in another intervention study .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2011-10; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Zager, MD, Study Chair — University New Mexico; Dana Miskulin, PhD, Principal Investigator — Tufts Medical Center; Jennifer Gassman, MD, Principal Investigator — The Cleveland Clinic; David Ploth, MD, Principal Investigator — Medical University of South Carolina; Manisha Jhamb, Principal Investigator — University of Pittsburgh; Mahboob Rahman, Principal Investigator — Case Western Reserve University
Locations (21):
- United States (21):
  - Dialysis Clinic Inc - Boston, Boston, Massachusetts
  - DaVita Boston, Boston, Massachusetts
  - Dialysis Clinic Inc - Walden Pond Clinic, Concord, Massachusetts
  - Dialysis Clinic Inc - Faulkner, Jamaica Plain, Massachusetts
  - Dialysis Clinic Inc - Somerville, Somerville, Massachusetts
  - Dialysis Clinic Inc - Albuquerque, Albuquerque, New Mexico
  - Dialysis Clinic Inc - Albuquerque South, Albuquerque, New Mexico
  - Dialysis Clinic Inc - Albuquerque East, Albuquerque, New Mexico
  - Dialysis Clinic Inc - Grants, Grants, New Mexico
  - Dialysis Clinic Inc - Rio Rancho, Rio Rancho, New Mexico
  - Centers for Dialysis Care East, Cleveland, Ohio
  - Centers for Dialysis Care - Shaker Heights, Cleveland, Ohio
  - Dialysis Clinic Inc - Oakland, Pittsburgh, Pennsylvania
  - Dialysis Clinic Inc - Banksville, Pittsburgh, Pennsylvania
  - Dialysis Clinic Inc - Point Breeze, Pittsburgh, Pennsylvania
  - Dialysis Clinic Inc - North Hills, Pittsburgh, Pennsylvania
  - Dialysis Clinic Inc - Magnolia Court, Charleston, South Carolina
  - Dialysis Clinic Inc - West Ashley, Charleston, South Carolina
  - Dialysis Clinic Inc - James Island, Charleston, South Carolina
  - Dialysis Clinic Inc - East Cooper, Mt. Pleasant, South Carolina
  - Dialysis Clinic Inc - Azalea Place, North Charleston, South Carolina

REFERENCES:
- [Derived] Miskulin DC, Gassman J, Schrader R, Gul A, Jhamb M, Ploth DW, Negrea L, Kwong RY, Levey AS, Singh AK, Harford A, Paine S, Kendrick C, Rahman M, Zager P. BP in Dialysis: Results of a Pilot Study. J Am Soc Nephrol. 2018 Jan;29(1):307-316. doi: 10.1681/ASN.2017020135. Epub 2017 Dec 6. PMID 29212839

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment to an Intensive BP Goal: Standardized predialysis systolic BP of 110-140 mmHg (intensive arm)
- Treatment to Standard BP Goal: Standardized predialysis systolic BP of 155-165 mmHg (standard arm)
Period: Overall Study
Arm/Group | Treatment to an Intensive BP Goal | Treatment to Standard BP Goal
Started | 62 | 64
Completed | 62 | 64
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment to an Intensive BP Goal: Treatment to a pre-dialysis standardized dialysis unit systolic blood pressure of 110-140 mm Hg
  Antihypertensive Agents: Study formulary consists of ACE/ARB, Beta Adrenergic Blocker, Calcium Channel Blocker, vasodilators, peripheral alpha antagonist and central alpha agonist.
  ACE I or ARB is first line, the order of addition of subsequent medications is per the discretion of the investigator
  Dry weight Challenge: Reduce the estimated dry weight of the patient's progressively over 2 -week intervals until the dry weight challenge is no longer tolerated or the patient is at BP goal
  Extend dialysis treatment time and re-challenge estimated dry weight: Extend dialysis treatment time and re-challenge estimated dry weight
- Treatment to Standard BP Goal: Treatment to a pre-dialysis Standardized dialysis unit systolic BP of 155-165 mm Hg
  Antihypertensive Agents: Study formulary consists of ACE/ARB, Beta Adrenergic Blocker, Calcium Channel Blocker, vasodilators, peripheral alpha antagonist and central alpha agonist.
  ACE I or ARB is first line, the order of addition of subsequent medications is per the discretion of the investigator
  Dry weight Challenge: Reduce the estimated dry weight of the patient's progressively over 2 -week intervals until the dry weight challenge is no longer tolerated or the patient is at BP goal
  Extend dialysis treatment time and re-challenge estimated dry weight: Extend dialysis treatment time and re-challenge estimated dry weight
- Total: Total of all reporting groups
Arm/Group | Treatment to an Intensive BP Goal | Treatment to Standard BP Goal | Total
Number analyzed (Participants) | 62 | 64 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (14.5) | 55 (10.8) | 56 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 25 | 55
  Male | 32 | 39 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 23 | 44
  Not Hispanic or Latino | 40 | 40 | 80
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 6
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 29 | 59
  White | 22 | 28 | 50
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 62 | 64 | 126

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Assessed for Intensive (110-140 mm Hg) and Standard (155-165mm Hg) Pre-dialysis Standardized BP Goal
Time Frame: one year
Measure: Number; unit: participants
Arm/Group | Treatment to an Intensive BP Goal | Treatment to Standard BP Goal
Number analyzed (Participants) | 62 | 64
participants | 62 | 64

2. Secondary Outcome: Number or Participants Assessed for Change in LV Mass
Time Frame: One year
Measure: Number; unit: participants
Arm/Group | Treatment to an Intensive BP Goal | Treatment to Standard BP Goal
Number analyzed (Participants) | 62 | 64
participants | 62 | 64

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Treatment to an Intensive BP Goal | Treatment to Standard BP Goal
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/64
Other Adverse Events (participants affected / at risk) | 0/62 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes